CLINICAL TRIAL: NCT06559137
Title: Prospective Evaluation of Post-operative Pain Management Using Peripheral Nerve Blocks in the Pediatric Population
Brief Title: Evaluation of Pain Management After Surgery When Using Nerve Blocks in the Pediatric Population
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2024-0774
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Sports Injuries in Children; Analgesia; Pain, Postoperative
Keywords: Narcotic use; Postoperative pain management; ACL reconstruction; Visual Analog Scale (VAS) pain scores; Multimodal pain management protocol
MeSH Terms: conditions — Lacerations; Agnosia; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomized after consent is obtained and will not know if they receive a single-shot peripheral nerve block. Due to current standard of care procedures, all patients will consent to receiving a peripheral nerve block despite their randomized group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peripheral Nerve Block (PNB) group (Active Comparator): * A 20 mL Adductor PNB will be injected where determined as best place by anesthesiologist
  * Patient will receive 0.2% plain Ropivacaine (perineural injection) regardless of weight
  * Patient will be given a purple surgical marker dot at/near the site of injection by the anesthesiologist
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- No Peripheral Nerve Block (PNB) group (No Intervention): - Patients will be given a purple surgical marker dot at/near the site where a PNB would be administered by the anesthesiologist, if they were randomized to the placebo group

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Patients who are randomized to the peripheral nerve block group will receive a pre-operative perineural injection of 0.2% plain Ropivacaine regardless of weight.
  Other Names: Naropin
  Arms: Peripheral Nerve Block (PNB) group

SUMMARY:
The goal of this randomized clinical trial is to determine if single-shot ropivacaine peripheral nerve blocks (PNB - perineural injections) for anterior cruciate ligament (ACL) reconstruction procedures in pediatric orthopaedic sports medicine patients provides significant pain relief and decreased narcotic use. The main questions it aims to answer are:

* Does ropivacaine significantly reduce Visual Analog Scale (VAS) pain scores and pain levels up to one week postoperatively?
* Does ropivacaine significantly decrease narcotic use (number of pills taken) up to one week postoperatively?

Researchers will compare the pain outcomes and narcotic use of participants who receive a single-shot ropivacaine peripheral nerve block to those of participants who do not receive a single-shot ropivacaine peripheral nerve block for their ACL reconstruction surgery. The goal is to understand if there is a significant difference in participant pain outcomes and narcotic use outside the first 24 hours postoperatively.

Participants will:

* receive either a single-shot ropivacaine peripheral nerve block intraoperatively or no peripheral nerve block during their ACL Quadriceps tendon graft or bone patellar tendon bone graft reconstruction surgery.
* receive and complete questionnaires at postoperative days 1, 4, and 7 regarding their pain scores, levels, and outcomes, effective pain treatments, overall pain interference, narcotic use (number of pills taken), and overall pain treatment satisfaction
* receive and complete secondary outcome measures of functional and psychological outcomes regarding their ACL reconstruction surgery at postoperative day 1

DETAILED DESCRIPTION:
This is a single institution, prospective, single-blinded (patient) randomized controlled trial to investigate the safety and pain-control efficacy and patient reported pain outcomes of PNBs in youth receiving ACLR. To be included, participants must be aged 13+ years at the time of surgery and present with an injury requiring an isolated ACL reconstruction with either a Bone-Patellar Tendon-Bone or Quadriceps tendon graft. Data will be collected from the patient's electronic medical record and from Oberd. Data collected will include age, height, weight, surgical information, diagnosis, and patient demographics. 160 participants (80 per treatment group) will be enrolled in the study with a minimum of 130 needed to complete the study.

As ACLR procedures are a frequent and standardized procedure at this institution, choosing to exclusively study this population offers a homogenous and plentiful sample. Pain protocols will follow a standard outline used by all participating surgeons to reduce variability between patients. The randomization technique of this study is supported by the equipoise of this institution's physicians regarding peripheral nerve blocks and the quantity of patients who this study's results will affect.

Patients will be approached pre-operatively for participation, after which the surgical team will be informed. Patients will be offered the choice to participate in the study and randomize their treatment group. If patients do not want their treatment to be randomized, they will not be included in the study. Data collection will involve the Wong-Baker Visual Analog Scale (VAS) and VAS 10-centimeter line 0-10 Numeric Pain Intensity Scale, and an institution specific pain questionnaire regarding analgesic medicine intake and complications daily from post-operative day one to post-operative day seven. Patients' medical records will also be reviewed for readmission, calls to their physician for pain, and other noted complications.

Patients will receive the following anesthesia doses by body weight (BW):

Pre-operatively:

* Regardless of age: 0.5 mg Midalozam per kg BW (intravenous, 15 mg maximum)
* If patient has history of PONV, 0.40 mg Emend per kg BW (pill), and 2 mg Midazolam (intravenous), and/or Scopolamine patch
* If patient has history of anxiety or PTSD, or exhibits anxiety symptoms before surgery:

0.1 mg Valium per kg BW (maximum 10 mg)

Intra-operatively:

* Amounts discretionary by patient vitals 0.5-1.0 mg Lidocaine per kg BW (intravenous -- no maximum) 3-4 mg Propofol per kg BW (no maximum) 1-2 mcg Fentanyl per kg BW (no maximum) 0.35 mg Ketamine per kg BW (no maximum) 0.1 mg Dexamethasone per kg BW (no maximum) If necessary: 0.004 - 0.006 mg Hydromorphone per kg BW (no maximum)
* Local Infiltration:

Regardless of weight: 10 mL Exparel and 20 mL 0.25% Marcaine - Optional: 10-20 mcg Dexmedetomidine per kg BW (for persistent tachycardia) <50% Nitrous If intubated/ventilated: 0.5-0.6 mg Rocuronium per kg BW, ~2 mg/kg Suggamadex for reversal If Tranexamic Acid administered: 15 mg per kg BW (10-15 min intravenous, maximum 1 g) For maintenance: 1 Minimum Alveolar Concentration (MAC) Sevoflurane and 15 mg Acetaminophen per kg BW (maximum 1 g) If necessary during emergence: 0.004-0.005 mg Hydropmorphone per kg BW, 0.5 mg Ketorolac per kg BW (maximum 30 mg), and 0.1 mg Ondansetron per kg BW (maximum 4 mg) If PACU medication required: 0.004-0.006 mg Hydromorphone per kg BW and 0.10- 0.15 mg Oxycodone per kg BW, and Metoclopramide, Dexamethasone, Promethazine, or Ondansetron

Peripheral Nerve Block Group Only:

* A 20 mL Adductor PNB will be injected where determined as best place by Anesthesiologist Patient will receive 0.2% plain Ropivacaine (perineural injection) regardless of weight
* Patient will be given a purple surgical marker dot at/near the site of injection by the anesthesiologist

Placebo Group Only:

- Patients will be given a purple surgical marker dot at/near the site where a PNB would be administered by the anesthesiologist, if they were randomized to the placebo group Modification / Update, MOD002-STU-2024-0774, Philip Wilson, 7/31/2025 STU-2024-0774, Wilson, FormA-Protocol, Mod_2, 07-31-25

Post-Operatively:

* Days 1-3: Alternate weight-adjusted Acetaminophen and 10 mg Ketorolac every 3 hours
* Days 4-7: Alternate weight-adjusted Acetaminophen and Ibuprofen every 3 hours
* Days 1-5: 40 mg Famotidine every 12 hours
* Rescue: Weight-adjusted Tramadol taken with Acetaminophen for severe pain (every 6 hours, maximum 8 doses) We will enroll 80 patients in each treatment group with 65 in each group needed for a sufficiently powered analysis. Patients will not be informed of their treatment group until after the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 13+ years at time of surgery
* Must present with injury requiring an ACLR procedure with a Bone Patellar Tendon Bone or Quadriceps graft
* Ability to provide assent, legally appointed representative available to provide informed consent

Exclusion Criteria:

* Patient <13 years old
* Requires fracture repair or another non-standardized surgery
* Any ACLR that requires the use of a graft type other than Bone Patellar Tendon Bone or Quadriceps tendon
* Any lower extremity procedure that is not primarily an ACLR
* Patient pregnancy
* Inability to provide assent or legally appointed representative to provide informed consent
* Prior history of hypersensitivity to Ropivacaine or any local anesthesia
* BMI ≥ 40

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Wong-Baker Face Pain Scale | Postoperative days 1, 4, and 7
  Scale with evocative faces from 0-10 (0 = No Pain, 10 = Worst Pain Possible) that assists children in communicating about their pain
Visual Analog Scale (VAS) 10-centimeter line 0-10 Numeric Pain Intensity Scale | Postoperative days 1, 4, and 7
  Sliding scale from 0-10 (0 = No Pain, 10 = Pain as bad as it could possibly be) that enables a more accurate estimate of pain score
Scottish Rite for Children-developed pain questionnaire | Postoperative days 1, 4, and 7
  Institutional questionnaire that asks how many narcotic pills the patient has taken (0 - 12 pills), if their pain is controlled, treatments that lessens their pain, term that best describes their pain, how much their pain has interfered with daily tasks and overall mood, and sleep interference due to pain.
Pain Management Patient Satisfaction questionnaire | Postoperative day 7
  Questionnaire that asks how satisfied patients are with their pain treatment (0 = Not Satisfied, 10 = Extremely Satisfied), if they contacted their physician due to ineffective pain treatment, how helpful the information provided for pain treatment was (0 = Not Helpful, 10 = Extremely Helpful), and a free response section to explain why they were not satisfied with their pain treatment and if they have any additional comments or suggestions based on their pain treatment.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Scale v1.0 - Global Health 7+2 | Preoperatively and within one week postoperatively.
  Questionnaire of outcomes regarding their overall health (scored 20-80, 20 = poor and 80 = good).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wilson, MD, Principal Investigator — Texas Scottish Rite Hospital for Children
Locations (1):
- Texas Scottish Rite Hospital for Children, Frisco, Texas, United States